CLINICAL TRIAL: NCT05133349
Title: A Prospective Phase II Efficacy and Safety Study of Anlotinib in Metastatic or Locally Advanced Pheochromocytoma/ Paraganglioma : Open-label Single-arm, Exploratory Trial.
Acronym: EASOAIPPGL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATPP
Record Dates: First submitted 2021-11-17; First posted 2021-11-24 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-09

CONDITIONS: Advanced or Metastatic Paraganglioma/ Pheochromocytoma
Keywords: Anlotinib; paraganglioma; pheochromocytoma
MeSH Terms: conditions — Paraganglioma; Pheochromocytoma | interventions — anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Anlotinib (Experimental): Anlotinib 12mg capsules given orally on once daily in 21-day cycle until disease progression or treatment intolerance(14 days on treatment from Day 1-14, 7 days off treatment from Day 15-21), the dose can be adjusted to 10mg or 8mg according to the specific conditions of the patient.
  Interventions: Drug: Anlotinib

INTERVENTIONS:
Drug: Anlotinib — Anlotinib 12mg capsules given orally on once daily in 21-day cycle until disease progression or treatment intolerance(14 days on treatment from Day 1-14, 7 days off treatment from Day 15-21), the dose can be adjusted to 10mg or 8mg according to the specific conditions of the patient.

SUMMARY:
This is an open-label phase II study of an investigational drug, anlotinib in participants with advanced malignant paraganglioma or pheochromocytoma. Pheochromocytoma and paraganglioma (PPGL) are tumors originating from the adrenal medulla or adrenal diplomatic sensory chain, respectively, which can synthesize and secrete large amounts of catecholamines. In this study, participants whose disease has advanced or spread despite prior standard therapy, will receive anlotinib for 2-weeks followed by a 1-week rest period, until disease progression (PD) or drug toxicity intolerance. Anlotinib is an investigational drug, which has been shown to shrink tumours in several tumour models. The study will evaluate the efficacy as well as the toxicity profile of anlotinib when used as an alternative treatment for participants with PPGL tumours.

DETAILED DESCRIPTION:
This study will be a single arm, open-label, phase II trial of anlotinib in participants with metastatic or locally advanced malignant pheochromocytoma or paraganglioma. Oral anlotinib (12 mg) will be administered to all participants daily for the first 2 weeks of a 3-week study cycle, followed by a 1 week rest. Participants will be assessed for response to study treatment using MRI/CT scans as well as bio-chemical tests, and will receive the study treatment for up to 12 months or until disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Participants with advanced, metastatic, recurrent or unresectable pheochromocytoma or paraganglioma. Pathology report or pathology slides (H&E) confirming histological diagnosis must be available at the time of enrollment.
* Must have measurable disease by RECIST v1.1.
* ECOG performance status 0-2, life expectancy of at least 6 months
* Adequate organ and marrow function was required (hemoglobin >= 8.0 g/dL (5.6 mmol/L); absolute neutrophil count (ANC) >= 1500/mm^3; platelet count >= 80,000/mm^3; creatinine =< 1.5 x ULN or creatinine clearance rate (CCr) ≥60ml/min, blood urea nitrogen (BUN) ≤2.5 × upper limit of normal (ULN); total bilirubin (TB) =< 1.5 X ULN; aspartate transaminase (AST) and alanine aminotransferase (ALT) <= 2.5 x ULN (if there are liver metastases, <= 5 x ULN); albumin (ALB) ≥25 g/L; urine protein/creatinine ratio =< 1 OR 24-hour urine protein < 1.5 gram)
* Blood pressure (BP) < 150 mmHg (systolic) and < 90 mmHg (diastolic); initiation or adjustment of BP medication is permitted prior to registration provided that the average of three BP readings at a visit prior to registration is < 150/90 mmHg; NOTE: all patients with secretory pheochromocytoma or paraganglioma are REQUIRED to: 1) be evaluated in consultation by a hypertension specialist with specific experience in the management of hypertension in the setting of catecholamine-secreting tumors (usually an endocrinologist, nephrologist, or a cardiologist), and in the setting of hormone-associated hypertension) receive alpha- and beta-adrenergic blockade for at least 7-14 days prior to initiation of anlotinib; the hypertension specialist of record for each patient should be committed to closely following the patient during the clinical study with evaluation by said specialist required at cycle 1 and 2 and thereafter on an as needed basis.
* Age greater or equal to 18 years old
* Participants who give a written informed consent obtained according to institutional guidelines
* Ability to complete questionnaire(s) by themselves or with assistance

Exclusion Criteria:

* Participants who have received bevacizumab, sunitinib, sorafenib, or pazopanib less than or equal to 2 weeks prior to starting study drug, or who have not recovered (grade 1) from the side effects of these therapies.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to anlotinib.
* Participants who have many influence factors toward oral medications
* Participants receiving concurrent treatment with other anti-cancer therapy chemotherapy/systemic therapy, radiotherapy, or immunotherapy =< 28 days prior to registration) given for paraganglioma or pheochromocytoma or failure to recover from toxicities. NOTE: concurrent therapy with octreotide is allowed providing that tumor progression on this therapy has been demonstrated; concurrent therapy with bisphosphonates (e.g. zoledronic acid) or denosumab is also allowed; There is no limit to the number of prior chemotherapy or biotherapy
* Participants with known untreated brain metastases are excluded. Participants having a history of brain metastasis that have been previously irradiated or resected greater than 3 months prior to enrollment and are clinically and radiographically stable will be considered for enrollment.
* Participants with another primary malignancy within 2 years prior to starting study drug, with the exception of adequately treated in-situ carcinoma of the uterine cervix, or skin cancer (such as basal cell carcinoma, squamous cell carcinoma, or non-melanomatous skin cancer)，also with the exception of other primary malignancy caused by related genetic diseases, such as VHL.
* Participants who have undergone major surgery (e.g. intra-thoracic, intra-abdominal or intra-pelvic), open biopsy or significant traumatic injury less than or equal to 4 weeks prior to starting study drug, or participants who have had minor procedures, percutaneous biopsies or placement of vascular access device 1 week prior to starting study drug, or who have not recovered from side effects of such procedure or injury
* Participants with any of the following concurrent severe and/or uncontrolled medical conditions which could compromise participation in the study (i.e. suffering from myocardial ischemia or above grade I myocardial infarction, arrhythmias and Class I heart failure; activity or failure to control severe infections; liver disease such as cirrhosis, decompensated liver disease, chronic active hepatitis; poorly controlled diabetes (FBG)>10mmol/L); urine protein≥++, etc.)
* Participants with any of the following conditions =< 6 months prior to registration: Cerebrovascular accident (CVA) or transient ischemic attack (TIA) Serious or unstable cardiac arrhythmia Admission for unstable angina or myocardial infarction Cardiac angioplasty or stenting Coronary artery bypass graft surgery Pulmonary embolism, untreated deep venous thrombosis (DVT) or DVT which has been treated with therapeutic anticoagulation =< 30 days Arterial thrombosis Symptomatic peripheral vascular disease
* Participants failed to heal wounds or fractures for Long-term
* Participants have HIV-positive or organ transplantation
* Pregnant or breastfeeding women or any subjects who refuse to use protocol required contraception
* Participants unwilling or unable to comply with the protocol
* Investigators consider that there are any conditions that may cause the participants to fail to perform study requirements.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-09-14 (Actual); Primary Completion 2023-09-14 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival Time | 2 years

SECONDARY OUTCOMES:
Overall response rate (PR) + (CR) | 2 years
Incidence of adverse events | 2 years
  Incidence of adverse events assessed by Common Terminology Criteria for Adverse safety profile of anlotinib

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Nanjing Medical Univerity, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No